CLINICAL TRIAL: NCT01165957
Title: A Comparison of Volumetric Wear Among DePuy Mobile and Fixed Bearing Knee Tibial Inserts
Brief Title: A Comparison of Wear Among Mobile and Fixed Bearing Knee Replacements
Status: Completed | Type: Observational
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, C. Anderson Engh, Jr., MD, Principal Investigator, Anderson Orthopaedic Research Institute
Other Study IDs: AORI2010-0102; Study #09010 (Other Grant/Funding Number: DePuy Orthopaedics, Inc.)
Record Dates: First submitted 2010-07-13; First posted 2010-07-20 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Osteoarthritis
Keywords: Knee replacement; Mobile and fixed bearings; Volumetric wear; Micro-CT analysis; Articular and backside wear
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mobile bearings: Tibial polyethylene inserts retrieved from total knee replacements where the insert is designed to slide or rotate on the metal baseplate.
- Fixed bearings: Tibial polyethylene inserts retrieved from total knee replacements where the insert is locked to the metal baseplate.

SUMMARY:
The purpose of this study is to determine the amount of polyethylene wear associated with knee replacement designs that incorporate either a fixed or mobile bearing. Tibial polyethylene inserts retrieved from modular total knee replacements during revision operations will be analyzed by obtaining micro-CT images of the retrieved inserts. The components of total volumetric polyethylene loss, including wear associated with the medial articular, lateral articular and backside regions of the insert be quantified by comparing the worn insert with an unworn control. The investigators hypothesize that the fixed bearing inserts where the polyethylene is locked to the metal baseplate will demonstrate more volumetric wear than the mobile bearing inserts that are designed to slide or rotate on the metal baseplate.

DETAILED DESCRIPTION:
Polyethylene wear is a major factor limiting the longevity of total knee arthroplasty. Evaluation of the volumetric wear of explanted polyethylene tibial inserts can provide valuable insight into the performance of different designs. Current technologies available to measure the volumetric wear of tibial inserts include gravimetric techniques, coordinate measuring machines (CMM), laser-scanning, and micro-CT.

In this study, we will employ micro-CT to determine volumetric wear because it allows us to obtain high-resolution three-dimensional images of the entire insert volume, including the surfaces as well as the interior of the insert. The micro-CT images will be used to reconstruct the entire three-dimensional geometry of the insert (including subsurface voids) and we will use image analysis software to partition the reconstructed insert into discrete regions (i.e. medial/lateral articulating surfaces, backside, and post), allowing us to determine how various regions contribute to total implant wear. By subdividing the insert into discrete regions, our analysis techniques will also enable us to account for material removed from the insert during explantation when evaluating implant wear. By comparing retrieved inserts with unworn controls using three-dimensional image analysis software, we will also quantify plastic deformation by measuring the volume of material that has deformed outside the confines of the control insert. Additionally, inspection of shape differences between the worn and unworn specimens will enable us to distinguish between implant wear, plastic deformation and volume differences associated with manufacturing tolerances. Although partial voluming effects can make edge detection challenging, high resolution micro-CT images tend to minimize these effects and we will use gravimetric measurements to determine an insert-specific Hounsfield threshold that will be used to define the image volume for each specimen. We will subsequently validate the accuracy of the reconstructed insert volume derived from the micro-CT image by comparing it with linear measurements from the actual specimen at several discrete locations.

The use of micro-CT scans to evaluate the in vivo volumetric wear associated with different designs will enable accurate measurement of volumetric polyethylene loss from different regions of the insert. This information will provide a better understanding of the clinical outcome associated with different design strategies and provide data to guide future development efforts. We hypothesize that fixed bearing inserts, where the polyethylene is locked to the metal baseplate, will demonstrate more volumetric wear than the mobile bearing inserts that are designed to slide or rotate on the metal baseplate.

Articular side wear will be measured by registering micro-CT images from retrieved and control inserts on unworn portions of the articular surface using the Analyze image analysis software (Mayo Biomedical Imaging Resource, Rochester, MN). Differences in volume among the retrieved and unworn control inserts will be evaluated accounting for plastic deformation that may occur in vivo. Volumetric wear for the entire insert and subregions will be calculated by subtracting the volume of plastic deformation (corresponding to regions of the retrieved insert outside the boundaries of the control insert) from the volume of material lost within the confines of the original insert geometry. We will compare wear among the mobile and fixed bearings using an Independent Sample t-test or Mann-Whitney U, depending on the distribution of the data. We will also use multiple linear regression analysis to examine the relationship between insert wear and other variables, including time in vivo, terminal sterilization technique for the insert and patient-related factors such as gender, age, and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* DePuy mobile and fixed bearing polyethylene tibial inserts retrieved after at least 12 months in vivo.
* Inserts terminally sterilized by gas plasma or with gamma radiation in oxygen-free barrier packaging.

Exclusion Criteria:

* Inserts that were sterilized by gamma radiation and exposed to oxygen in packaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrieved polyethylene tibial inserts archived as part the Anderson Orthopaedic Research Institute's implant retrieval program.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Total Volumetric Wear | At time of revision (average 46 months)
  Total volumetric polyethylene wear will be measured among mobile and fixed bearing tibial inserts retrieved during a revision surgery.

SECONDARY OUTCOMES:
Local Volumetric Wear | At time of revision (average 46 months)
  Wear from different regions, including the medial articular, lateral articular and backside surfaces, will be evaluated. Maximum linear penetration will also be determined for the medial and lateral compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Hopper, Jr., PhD, Study Director — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States

REFERENCES:
- [Background] McEwen HM, Barnett PI, Bell CJ, Farrar R, Auger DD, Stone MH, Fisher J. The influence of design, materials and kinematics on the in vitro wear of total knee replacements. J Biomech. 2005 Feb;38(2):357-65. doi: 10.1016/j.jbiomech.2004.02.015. PMID 15598464
- [Background] Jennings LM, Bell CI, Ingham E, Komistek RD, Stone MH, Fisher J. The influence of femoral condylar lift-off on the wear of artificial knee joints. Proc Inst Mech Eng H. 2007 Apr;221(3):305-14. doi: 10.1243/09544119JEIM215. PMID 17539585
- See also: Website for Anderson Orthopaedic Research Institute — http://aori.org